CLINICAL TRIAL: NCT03250338
Title: Phase III Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy of the Addition of Crenolanib to Salvage Chemotherapy Versus Salvage Chemotherapy Alone in Subjects ≤ 75 Years of Age With Relapsed/Refractory FLT3 Mutated Acute Myeloid Leukemia
Brief Title: Study Investigating the Efficacy of Crenolanib With Chemotherapy vs Chemotherapy Alone in R/R FLT3 Mutated AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARO-013; 2017-001600-29 (EudraCT Number)
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia With FLT3 Activating Mutations
MeSH Terms: conditions — Recurrence | interventions — crenolanib; Cytarabine; Mitoxantrone; fludarabine; Idarubicin; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crenolanib (Experimental): Crenolanib following salvage chemotherapy
  Interventions: Drug: Crenolanib; Drug: Cytarabine; Drug: Mitoxantrone; Drug: Fludarabine; Drug: Idarubicin; Drug: G-CSF
- Placebo (Placebo Comparator): Placebo following salvage chemotherapy
  Interventions: Drug: Cytarabine; Drug: Mitoxantrone; Drug: Placebo Oral Tablet; Drug: Fludarabine; Drug: Idarubicin; Drug: G-CSF

INTERVENTIONS:
Drug: Crenolanib — Crenolanib will be administered orally
  Other Names: Crenolanib besylate
  Arms: Crenolanib
Drug: Cytarabine — HAM regimen
  FLAG-Ida
Drug: Mitoxantrone — HAM regimen
Drug: Placebo Oral Tablet — Placebo will be administered orally
  Arms: Placebo
Drug: Fludarabine — FLAG-Ida regimen
Drug: Idarubicin — FLAG-Ida regimen
Drug: G-CSF — FLAG-Ida regimen

SUMMARY:
This is a randomized, multi-center, double-blind, placebo-controlled study designed to evaluate the efficacy of crenolanib administered following salvage chemotherapy, consolidation chemotherapy, post bone marrow transplantation and as maintenance in relapsed/refractory AML subjects with FLT3 activating mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of AML according to World Health Organization (WHO) 2016 classification
2. Presence of FLT3-ITD and/or D835 mutation(s)
3. Subjects must be primary refractory or relapsed to 1st line intensive treatment for AML or refractory or relapsed after second line of treatment for AML
4. Age ≥ 18 years and ≤ 75 years
5. Adequate hepatic function
6. Adequate renal functions
7. ECOG performance status ≤ 3

Exclusion Criteria:

1. Known clinically active central nervous system(CNS) leukemia
2. Severe liver disease
3. Known, active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
4. Prior anti-leukemia therapy within the 14 days prior to randomization. Prior use of quizartinib or gilteritinib must be discontinued 21 days prior to randomization. Prior use of hydroxyurea or other palliative treatment for leukocytosis is allowed.
5. Previous treatment with crenolanib or prior participation in clinical trial involving crenolanib.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 3 years

SECONDARY OUTCOMES:
Overall Survival | 3 years
Relapse-free Survival (RFS) | 3 years
Complete remission rate (CR) | 3 years
MRD negative complete remission rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Wang, MD, Principal Investigator — Roswell Park Cancer Institute, Buffalo, New York, United States, 14263
Locations (62):
- United States (9):
  - City of Hope National Medical Center, Sacramento, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Kansas University, Kansas City, Kansas
  - Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
- University of Alberta, Edmonton, Alberta, Canada
- France (12):
  - Hospital Avicenne, Bobigny
  - CHU Grenoble Alpes, Grenoble
  - Hospital Center of Versailles (Le Chesnay), Le Chesnay
  - Hospital Claude Huriez - Chru Lille, Lille
  - Institut Paoli-Calmettes, Marseille
  - CHU de Nantes - Hôtel Dieu, Nantes
  - University Hospital Nice L'Archet, Nice
  - Hôpital St Louis, Paris
  - CHU de Bordeaux, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Institut Universitaire du Cancer Toulouse, Toulouse
- Germany (6):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Essen (AöR), Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Münster, Münster
- Italy (19):
  - Policlinico Tor Vergata, Roma, RM
  - AOU Policlinico Sant'Orsola-Malpighi, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - AOU Careggi, Florence
  - IRST - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - IRCCS San Raffaele Hospital, Milan
  - IRCCS Foundation Ca 'Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Europeo di Oncologia, Milan
  - Aorn Antonio Cardarelli, Napoli
  - AOU Federico II, Napoli
  - AOU Maggiore della Carità, Novara
  - AO Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - AO Ospedali Riuniti Marche Nord, Pesaro
  - Ospedale Santa Maria delle Croci di Ravenna, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - AO Ordine Mauriziano di Torino, Torino
  - Policlinico GB Rossi, University Hospital Verona, Verona
  - AULSS n 8 Berica Ospedale San Bortolo, Vicenza
- Spain (15):
  - Hospital U. Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Central de Asturias (HUCA), Oviedo, Principality of Asturias
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - San Pedro de Alcantara Hospital, Cáceres
  - Reina Sofia University Hospital, Córdoba
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Gregorio Maranon Servicio de Hematologia y Hemoterapia, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital U. Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario y Politecnico La Fe, Valencia